CLINICAL TRIAL: NCT03261375
Title: Prospective Multicenter Randomized Parallel Controlled Clinical Trial to Evaluate the Safety and Effectiveness of a Radiofrequency Renal Denervation System for the Treatment of Essential Hypertension
Brief Title: To Evaluate Safety and Efficacy of a Radiofrequency Renal Denervation System in Treatment of Essential Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Golden Leaf MedTec Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MLWY-SXX201601
Record Dates: First submitted 2017-08-21; First posted 2017-08-25 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Hypertension
Keywords: Hypertension; Renal Denervation
MeSH Terms: conditions — Hypertension | interventions — Radionuclide Generators; Catheters; Antihypertensive Agents; Nifedipine; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Both patients and site investigators who evaluate the patients were blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renal denervation (RDN) Group (Experimental): Receive standardized 2 drugs (Nifedipine and hydrochlorothiazide) treatment and renal denervation treatments (RDN)
  Interventions: Device: Renal Artery Radiofrequency Ablation System (Generator and Catheter ); Drug: Antihypertensive Agents
- Control Group (Sham Comparator): Receive standardized 2 drugs (Nifedipine and hydrochlorothiazide) treatment and renal artery angiography only
  Interventions: Drug: Antihypertensive Agents; Device: Sham Procedure

INTERVENTIONS:
Device: Renal Artery Radiofrequency Ablation System (Generator and Catheter ) — A renal denervation system with a mesh 6-electrode radiofrequency ablation catheter and multi-channel radiofrequency generator
  Arms: Renal denervation (RDN) Group
Drug: Antihypertensive Agents — Calcium channel blocker, Diuretic
  Other Names: Nifedipine and hydrochlorothiazide
Device: Sham Procedure — Catheterization without renal denervation
  Arms: Control Group

SUMMARY:
This is a prospective, multicenter, randomized sham-controlled trial to evaluate safety and efficacy of a multi-electrode radiofrequency renal denervation system (Netrod® System) in treating patients with uncontrolled essential hypertension.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized sham-controlled trial. Patients with uncontrolled hypertension (office BP ≥150/90 and <180/110mmHg, and average SBP ≥135mmHg by 24-hour ambulatory BP monitoring (ABPM), after taking ≥2 antihypertensive drugs with stable dose for ≥ 4 weeks) were screened after informed consent. All eligible patients first entered a lead-in period for ≥4 weeks of standardized medication (Nifedipine + hydrochlorothiazide), and those continued to meet definition of uncontrolled hypertension were randomized 2:1 to RDN group and sham control group (renal artery angiography only). All continued with the 2-drug regimen and were evaluated at 7, 30, 60, 90 and 180 days post procedure. Both patients and site investigators who evaluate the patients were blinded to treatment assignment. The primary endpoint is office SBP change from baseline at 6 months post procedure. Secondary endpoints include changes from baseline of office DBP. 24-hour ABPM at 6 months post procedure and safety events.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with age of 18 to 65 years old (include 65), male or female;
2. Subject with essential hypertension who has an office BP of ≥150/90mmHg and <180/110 mmHg (both SBP and DBP meet the criteria), and an average SBP of ≥ 135mmHg measured by 24-hour ABPM, after taking ≥ 2 antihypertensive medications for ≥ 4 weeks;
3. Subject with the resting heart rate ≥70bpm, if not taking beta-blockers (this criterion does not apply to those taking beta-blockers);
4. Subject with confirmed diagnosis of essential hypertension;
5. Subject with or without accessary renal arteries;
6. Subject who has signed the informed consent form, agrees to participate in this clinical trial, and is willing to comply with the required follow-ups per the trial protocol.

Exclusion Criteria:

1. Subject who is pregnant, nursing or planning to become pregnant during the study;
2. Subject with the shape and structure of unilateral or bilateral renal artery that are not suitable for ablation procedure (renal artery stenosis more than 50%, renal aneurysm, renal artery abnormality, renal artery diameter <4mm or treatable segment length <20mm);
3. Subject who has unilateral kidney or kidney transplant;
4. Subject with a history of renal artery interventional therapy or renal denervation;
5. Subject with any conditions that may affect the accuracy of blood pressure measurement: such as the diameter of the upper arm is too large relative to the cuff, arrhythmia;
6. Subject with secondary hypertension;
7. Subject with pseudo-hypertension;
8. Subject with orthostatic hypotension;
9. Subject with eGFR <45mL/min/l.73m2;
10. Subject with average SBP is < 135mmHg on 24-hour ABPM;
11. Subject with a history of hospitalization for hypertensive emergency within past one year;
12. Subject with type I diabetes mellitus;
13. Subject with primary pulmonary hypertension;
14. Subject with a history of bleeding diathesis and hematological disorders;
15. Subject with a history of embolism within past 6 months;
16. Subject with a history of acute coronary syndrome within past 6 months;
17. Subject with a history of ventricular fibrillation, polymorphic ventricular tachycardia within past 6 months;
18. Subject with serum HIV-positive;
19. Subject who is allergic to contrast agents;
20. Subject with mental illness or any psychological problems that may interfere with the participating in the study;
21. Subject with a history of stroke or transient ischemic attack (TIA) within past 3 months;
22. Subject with malignant tumors or end-stage disease;
23. Subject with severe peripheral vascular disease or abdominal aortic aneurysm;
24. Subject with severe heart valve stenosis;
25. Subject with cardiac insufficiency (NYHA class III~IV);
26. Subject with hyperthyroidism or hypothyroidism;
27. Subject with severe electrolyte or liver function abnormalities;
28. Subject who requires mechanical ventilation other than nocturnal respiratory support for sleep apnea;
29. Subject with acute or severe systemic infection;
30. Subject with a history of pacemaker implantation;
31. Subject with a history of major surgery or trauma within 30 days prior to enrollment;
32. Subject who has planned surgery or cardiovascular intervention within the next 6 months;
33. Subject who is participating in other drug or medical device clinical trials;
34. Subject who has known drug or alcohol dependence, difficulty to understand the trial protocol, inability/unwillingness to follow the trial protocol;
35. Subject who is unsuitable for participating in this study in the opinion of investigators;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2022-12-26 (Actual)

PRIMARY OUTCOMES:
Office SBP change from baseline at 6 months post procedure | From baseline to 6 months
  Change in office blood systolic pressure (SBP) at 6 months post procedure

SECONDARY OUTCOMES:
Office DBP change from baseline at 6 months post procedure | From baseline to 6 months
  Change in office blood diastolic pressure (DBP) at 6 months post procedure
Changes in 24-hour ambulatory BP at 6 months post procedure | From baseline to 6 months
  Changes in 24-hour ambulatory SBP and DBP from baseline at 6 months post procedure measured by 24-hour ABPM
Incidence of achieving target office SBP (90mmHg≤SBP<140mmHg) at 6 months post procedure | From baseline to 6 months
  Patient proportion of achieving target office SBP (90mmHg≤SBP<140mmHg) at 6 months post index procedure
Proportion of office SBP decreased by ≥ 5mmHg at 6 months post index procedure | From baseline to 6 months
  Proportion of office SBP decreased by ≥ 5mmHg at 6 months post index procedure
The rate of major adverse events (MAE) through 6 months post index procedure | From index procedure to 6 months post procedure
  The rate of major adverse events (MAE) through 6 months post index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Yujie Zhou, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (25):
- China (25):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Shijiazhuang People's Hospital, Shijiazhuang, Hebei
  - Nanyang Second People's Hospital, Nanyang, Henan
  - The Seventh People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The 1st Affiliated Hospital Zhengzhou University, Zhengzhou, Henan
  - Zhongda Hospital, Southeast University, Nanjing, Jiangsu
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Heze Municipal Hospital, Heze, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The First People's Hospital of Jining, Shandong Province, Jining, Shandong
  - Qingdao Central Hospital, Qingdao, Shangdong
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Tangdu Hospital, Fourth Military Medical University, Xi’an, Shanxi
  - Xianyang Hospital of Yan 'an University, Yanan, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Huaxi Hospital, Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Xinjiang Autonomous Region People's Hospital, Ürümqi, Xinjiang
  - Run Run Shaw Hospital, Zhejiang University School of Medicine, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No